CLINICAL TRIAL: NCT04056312
Title: A Randomized Clinical Trial Examining The Efficacy of The Group Administered Modified Story Memory Technique (mSMT) in Persons With TBI
Brief Title: Modified Story Memory Technique (mSMT) in Persons With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director NNL & TBI, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-926-16
Record Dates: First submitted 2017-08-15; First posted 2019-08-14 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Traumatic Brain Injury
Keywords: memory; learning; cognition; traumatic brain injury; treatment and therapy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group memory retraining (Experimental): Experimental group will be receiving memory retraining exercises via lap top twice a week for 5 weeks. Four people in a group.
  Interventions: Behavioral: Group Memory retraining exercises
- Placebo (Placebo Comparator): Experimental group will be receiving memory retraining exercises via lap top twice a week for 5 weeks. Four people in a group.
  Interventions: Behavioral: Placebo controlled group memory exercise training

INTERVENTIONS:
Behavioral: Group Memory retraining exercises — Experimental group will be receiving memory retraining exercises via lap top twice a week for 5 weeks. Four people in a group.
  Arms: Group memory retraining
Behavioral: Placebo controlled group memory exercise training — Placebo group will be receiving memory retraining exercises via lap top twice a week for 5 weeks. Four people in a group.
  Arms: Placebo

SUMMARY:
The current RCT is designed to:

1. test the efficacy of the group based mSMT in persons with TBI on NPE, the current gold-standard for measuring memory functioning
2. assess the effectiveness of the group mSMT on more global measures of everyday life, including an objective measure shown through our previous work to be sensitive to memory changes following the mSMT, as well as additional questionnaires to be completed by both the participant and a significant other
3. evaluate the changes in brain functioning following treatment with the mSMT via fMRI and
4. evaluate the long-term effects of the treatment protocol.

To accomplish these goals investigators will conduct a double-blind, placebo-controlled, RCT, applying the group mSMT to a sample of 60 participants with moderate to severe TBI (30 treatment; 30 control).

DETAILED DESCRIPTION:
Outcome measures will assess objective memory abilities, everyday memory abilities and patterns of cerebral activation during learning. A long-term follow-up assessment will be conducted, designed to measure the impact of the mSMT 3 months following treatment completion. Alternate forms will be utilized wherever available.

ELIGIBILITY:
Inclusion Criteria:

* I am between the ages of 18-65.
* I have had a Traumatic Brain Injury at least one year ago.
* I can read and speak English fluently.
* I have difficulties with learning and memory skills.

Exclusion Criteria:

* I am currently taking steroids and /or benzodiazepines as determined by study staff review of my medications.
* I have had a prior stroke or neurological injury/disease other than a traumatic brain injury.
* I have a history of significant psychiatric illness (for example, bipolar disorder or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II.
* I have unstable or uncontrolled seizures.
* I have a significant alcohol or drug abuse history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test | Change will be assessed. Scales will be administered at 3 time points;pretreatment immediately following 5 months later
  Change on scores on memory tests will be assessed using the California Verbal Learning Test
The Traumatic Brain Injury-Quality of Life Scale | Change will be assessed. Scales will be administered at 3 time points;pretreatment immediately following 5 months later
  Self-reports of emotional functioning, memory functioning and quality of life on The Traumatic Brain Injury-Quality of Life Scale, which measures these constructs. DVs will be change on the Depression subscale (range: 0-40; lower score is better) and Cognition scale (range: 0-40; higher score is better).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Green, PhD, Study Chair — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States